CLINICAL TRIAL: NCT02065362
Title: Administration Of TGF-beta Resistant Cytotoxic T-Lymphocytes to Patients With EBV-positive Nasopharyngeal Carcinoma (RESIST-NPC)
Brief Title: TGF-beta Resistant Cytotoxic T-lymphocytes in Treatment of EBV-positive Nasopharyngeal Carcinoma / RESIST-NPC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Helen Heslop, Director CAGT, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33954: RESIST-NPC; P01CA094237 (NIH)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: EBV-positive Nasopharyngeal Carcinoma
Keywords: EBV positive; TGFbeta; Nasopharyngeal carcinoma; cytotoxic T lymphocytes
MeSH Terms: conditions — Camurati-Engelmann Syndrome; Nasopharyngeal Carcinoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DNR.NPC-specific T cells or DNR.NPC-specific T cells + c/f (Experimental): DNR.NPC-specific T cells or DNR.NPC-specific T cells + c/f
  Interventions: Biological: DNR.NPC-specific T cells; Biological: DNR.NPC-specific T cells + cyclophosphamide + fludarabine

INTERVENTIONS:
Biological: DNR.NPC-specific T cells — Each patient will receive 2 infusions, 14 days apart, according to the following dosing schedule:
  Dose Level 1:
  Day 0: 2 x 10^7 cells/m^2
  Day 14: 2 x 10^7 cells/m^2
  The doses are calculated according to the total T cell number.
Biological: DNR.NPC-specific T cells + cyclophosphamide + fludarabine — Patients will receive cyclophosphamide and fludarabine for 3 days before receiving the DNR.NPC-specific T cells.
  Each patient will receive infusions according to the following dosing schedule:
  Dose Level 2:
  Cy/Flu on Days -4 to -2 and then 4 x 10^7 cells/m^2 on Day 0, Day 1 or Day 2
  Dose Level 3:
  Cy/Flu on Days -4 to -2 and then 1 x 10^8 cells/m^2 on Day 0, Day 1, or Day 2

SUMMARY:
Patients have nasopharyngeal carcinoma (NPC). This study is a gene transfer research study using special immune cells.

Most patients with NPC show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of almost all patients with advanced stage NPC, suggesting that it may play a role in causing the disease. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called T cells, that have been trained to recognize and kill special parts of EBV infected cells can survive in patient's blood and affect the tumor.

We already have given EBV-specific cytotoxic T cells to 30 patients with active NPC and have seen anti-tumor activity in 14 of 30 patients. We are now trying to find out if we can improve this treatment.

First, we want to give T cells where more of the cells recognize at least two of the four EBV proteins expressed on NPC cells. We call these cells NPC-specific cytotoxic T cells.

Second, we found that T cells work better if we add a receptor to the T cells called DNR (Dominant Negative Receptor). DNR makes T cells resistant to TGFbeta, a factor secreted by cancer cells that helps them escape being killed by the immune system. In this study we will therefore place the DNR gene into NPC-specific T cells (DNR.NPC-specific T cells).

In other clinical studies using T cells, some investigators found that giving chemotherapy before the T cell infusion can improve the amount of time the T cells stay in the body and therefore the effect the T cells can have. Giving chemotherapy before a T cell infusion is called lymphodepletion since the chemotherapy is specifically chosen to decrease the number of lymphocytes in the body. Decreasing the number of patient's lymphocytes first should allow the T cells we infuse to expand and stay longer in their body, and potentially kill cancer cells more effectively.

The chemotherapy we will use for lymphodepletion is a combination of cyclophosphamide and fludarabine. Cyclophosphamide and fludarabine are the chemotherapy agents most commonly used for lymphodepletion in immunotherapy clinical trials.

DETAILED DESCRIPTION:
Blood will be collected from the patient to make LMP/BARF1/EBNA1 (NPC)-specific T cells. To grow NPC-specific T cells we have to use special cells called antigen-presenting cells, which train the patient's T cells to be NPC specific. Antigen presenting cells, so called monocytes or dendritic cells, will be grown/isolated from the patient's blood. In addition, we use a cell line called K562 as antigen-presenting cells that has had genes put inside it, which encourage the patient's T cells to grow. K562 cells are cancer cells. As such, if injected they could cause cancer. The cells have been treated with radiation so they cannot grow.

These antigen-presenting cells are coated with a specially produced mixture of LMP, EBNA1 and BARF protein fragments called peptides. These coated antigen-presenting cells are then used to generate the patient's NPC-specific T cells in the presence of growth factors. To get the DNR to attach to the surface of these NPC-specific T Cells, we also inserted the DNR gene into the NPC-specific T cells (DNR.NPC-specific T cells). This is done with a virus called a retrovirus that has been made for this study. This virus will carry the DNR gene into the cells.

Once we have made sufficient numbers of DNR.NPC-specific T cells we will freeze the cells and test them to make sure they recognize EBV proteins present in NPC.

Patients will get treated with 1) either two doses of DNR.NPC-specific T cells (the second dose will be given 2 weeks after the first dose) or 2)cyclophosphamide and fludarabine for 3 days before receiving the DNR.NPC-specific T cells.

The cyclophosphamide and fludarabine will be given through a needle inserted into a vein or patient's port-a-cath).

The T cells will be thawed and infused through a central line, or through a vein in the patient's arm over 1 to 10 minutes. Patients will be followed in the clinic after the infusion for 1 to 4 hours.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

Medical tests before treatment:

Before being treated, the patient will receive a series of standard medical tests:

Physical exam Imaging Study Blood tests to measure blood cells, kidney and liver function Measurements of the tumor by routine imaging studies. We will use the imaging study that was used before to follow the patient's tumor: Computer Tomogram (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET/CT)

Medical tests during and after treatment:

The patient will receive standard medical tests when they are getting the infusions and after:

Physical exams Blood tests to measure blood cells, kidney and liver function Imaging study 8 weeks after the 1st T-cell infusion(for patients receiving only DNR.NPC-specific T cells ) or Imaging study 6 weeks after the T-cell infusion (for patients receiving fludarabine and cyclophosphamide before DNR.NPC-specific T-cell infusion).

To learn more about the way the DNR.NPC-specific T cells are working and how long they last in the body, an extra 60ml or 3ml/kg of body weight of blood (whichever is less) will be taken pre-chemotherapy (for the patients receiving chemotherapy), on the day of the T-cell infusion (before and at the end of the T-cell infusion), 1, 2, 3, 4. 6, and 8 weeks( the last time point only for patients receiving DNR.NPC-specific T-cells only) after the T-cell infusion and every 3 months for 1 year, every 6 months for 4 years, then yearly for a total of 15 years. One additional blood sample might be drawn 3 to 4 days post the 1st T-cell infusion; this is optional. This volume is considered safe, but may be decreased if the patient is anemic. In addition to the blood tests, the patient will receive 2 imaging studies as stated above.

During the time points listed above, if the DNR.NPC-specific T cells are found in patient's blood at a certain amount an extra 5ml of blood may need to be collected for additional testing.

ELIGIBILITY:
Inclusion Criteria:

The patient must meet the following eligibility inclusion criteria at the time of PROCUREMENT:

* Nasopharyngeal Carcinoma in first or subsequent relapse or with primary refractory disease
* EBV positive tumor
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

The patient must meet the following eligibility criteria to be included for TREATMENT:

* Nasopharyngeal Carcinoma in first or subsequent relapse or with primary refractory disease
* EBV positive tumor
* Patients with life expectancy greater than or equal to 6 weeks
* Bilirubin less than or equal to 3x upper limit of normal
* AST less than or equal to 5x upper limit of normal
* ANC>750/microliter
* Platelets > 50,000/microliter
* Hgb ≥ 7.0g/dl (can be transfused)
* Creatinine less than or equal to 2x upper limit of normal for age, Creatinine clearance (as estimated by Cockcroft Gault or Schwartz) greater than or equal to 60 ml/min
* Pulse oximetry of > 90% on room air
* Off investigational therapy for 4 weeks prior to study entry
* Karnofsky or Lansky score of greater than or equal to 50%
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

At time of Procurement:

•Known HIV positivity

At time of Treatment:

* Pregnant or lactating
* Severe intercurrent infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a dose limiting toxicity | 8 weeks
  Determine the safety of escalating doses of intravenous infusions of autologous TGFbeta-resistant NPC-specific cytotoxic T-lymphocytes with lymphodepleting chemotherapy for dose levels 2 and 3 in patients with EBV-positive nasopharyngeal carcinoma (NPC).

SECONDARY OUTCOMES:
Amount of T cells in the blood after the infusions | 15 years
  Determine the survival and the immune function of TGFbeta-resistant NPC specific T cells.

OTHER OUTCOMES:
Number of patients with a response to the T cells | 8 weeks
  Assess the anti-viral and anti-tumor effects of TGFbeta-resistant NPC specific T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine/Texas Children's Hospital /Houston Methodist Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT02065362/ICF_000.pdf